CLINICAL TRIAL: NCT02389530
Title: Use of Fluorescein Dye for the Removal of Brain Tumors
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO14100616
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2017-11

CONDITIONS: Brain Neoplasms
Keywords: glioma; neoplasms
MeSH Terms: conditions — Brain Neoplasms; Glioma; Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- interventional group: All participants will receive the study intervention, intravenous administration of fluorescein dye prior to brain tumor removal.
  Interventions: Drug: Fluorescein

INTERVENTIONS:
Drug: Fluorescein — Fluorescein will be administered intravenously at a dose between 250 mg and 400 mg in the experimental arm.

SUMMARY:
Fluorescein is a dye agent that can be injected through an intravenous line. It has been shown to help tell the difference between brain tumor tissue and normal brain tissue when it is used together with a specialized filter on a microscope in the operating room. The investigators plan to study the use of fluorescein in the removal of brain tumors at a low dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 or greater
2. Plan for elective removal of a brain tumor at UPMC Shadyside with either Dr. Engh or Dr. Amankulor.

Exclusion Criteria:

1. History of adverse reaction to fluorescein.
2. Emergent surgical procedure (consent not feasible).
3. Creatinine of > 2.0 (drug is excreted renally).
4. Known ongoing pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or above pending elective removal of an intraparenchymal brain tumor.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Adverse event assessment | 3 years
  Assessment of frequency of adverse events related to fluorescein administration, especially anaphylaxis

SECONDARY OUTCOMES:
Degree of tumoral resection | 3 years
  Volumetric assessment of amount of tumor removed, compared to historical controls
Clinical status after surgery | 3 years
  Assessment of new deficit in speech, motor function, sensation or vision based on post-operative neurological examination: NIH stroke scale scores will be measured for all participants pre- and post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan Engh, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States